CLINICAL TRIAL: NCT02705729
Title: Clinical Performance of a Newly Developed Glass Ionomer Restorative Material for Posterior Restorations in an Adolescent Population
Brief Title: Clinical Performance of Posterior Glass Ionomer Restorations in Adolescents (KETAC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: 3M Oral Care (Other)
Responsible Party: Principal Investigator, Suzanne E Fournier, Clinical Assistant Professor and Postgraduate Program Director, Louisiana State University Health Sciences Center in New Orleans
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LSUHSC-NO #9270
Record Dates: First submitted 2016-03-07; First posted 2016-03-10 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Dental Caries
Keywords: dental caries; proximal surfaces; posterior teeth; carious lesions; tooth diseases; dental restorations; glass-ionomer
MeSH Terms: conditions — Dental Caries; Tooth Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketac Universal (Active Comparator): Simplified glass ionomer tooth filling
  Interventions: Device: Ketac Universal
- Ketac Molar Quick (Active Comparator): Glass ionomer tooth filling
  Interventions: Device: Ketac Molar Quick

INTERVENTIONS:
Device: Ketac Universal — High-viscous glass ionomer restorative material used as posterior dental filling. This material does not require a dentin conditioning step.
  Other Names: Ketac Universal Aplicap Glass Ionomer Restorative
  Arms: Ketac Universal
Device: Ketac Molar Quick — High-viscous glass ionomer restorative material used as posterior dental filling. This material requires a dentin conditioning step.
  Other Names: Ketac Molar Quick Aplicap Glass Ionomer Restorative
  Arms: Ketac Molar Quick

SUMMARY:
The purpose of this study is to determine whether two tooth-colored glass ionomer materials are effective for load-bearing dental fillings.

DETAILED DESCRIPTION:
In this post-market longitudinal prospective randomized control clinical trial, posterior class II restorations will be evaluated for their clinical performance. The study will investigate the efficacy of two high-strength glass ionomer restorative materials for a period of up to 3 years.

ELIGIBILITY:
Criteria:

* Inclusion Criteria:
* needs 2 Class II posterior restorations
* in good health
* sufficient oral hygiene
* vital tooth
* caries in the outer and/or middle third of dentin
* teeth must have at least one proximal contact to be restored
* isthmus is less than half the intercuspal distance
* has one or more enamel-supported antagonistic contact.
* both study restorations are not in contact with each other

Exclusion Criteria:

* pregnant or breast feeding
* erosion/eating disorders
* bruxism/traumatic malocclusion
* pulpitis
* cusp replacement
* radiographic bone loss/increased tooth mobility

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-08-03; Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Restoration survival | 3 years
  Survival based on criteria for posterior glass ionomer restorations

SECONDARY OUTCOMES:
Clinical Performance of restoration and restored tooth | 3 years
  Clinical performance based on criteria for posterior glass ionomer restorations
Additional Collection of Adverse Events Data | 3 years
  Data collection of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde C Peters, DMD, PhD, Study Director — LSUHSC School of Dentistry
Locations (1):
- Lousiana State University Health Science Center, School of Dentistry, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided